CLINICAL TRIAL: NCT05658614
Title: Evaluation of Immunogenicity and Safety of a New Vaccine Schedule Using the Vaccine Candidate Sm14 Against Schistosomiasis in Adults With a History of S. Mansoni and / or S. Haematobium Infection.
Brief Title: Anti-Schistosomiasis Sm14-vaccine in Senegal
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, MIRIAM TENDLER, MD, PhD, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sm14-2c-Sn
Record Dates: First submitted 2021-11-10; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Schistosomiasis Mansoni; Schistosomiasis Haematobium; Vaccination; Infection
MeSH Terms: conditions — Schistosomiasis mansoni; Schistosomiasis haematobia; Infections

STUDY DESIGN:
Intervention Model Description: Main objective: to compare the immunological quality of the new vaccination schedule (amplitude and duration) versus the vaccination schedule used in the previous trials, by studying the Sm14 specific antibody response induced both quantitatively and qualitatively. The hypothesis is to obtain a mean response quantitatively higher with the new vaccine schedule.
  Secondary objective: safety profile of the two vaccine schedules studied.
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Group Vacc3) (Active Comparator): Volunteers will receive three (3) intramuscular injections into the deltoid muscle of 0.5mL of of the Sm14+ GLA-SE vaccine on D0, W4 and W8. (D = Day; W = Week). (Vaccination schedule used in previous phases).
  Interventions: Biological: Sm14 recombinant vaccine+ GLA-SE adjuvant
- Arm 2 (Group Vacc2+1) (Experimental): Volunteers will receive three (3) intramuscular injections of the Sm14+ GLA-SE vaccine into the deltoid muscle of 0.5mL of vaccine on D0, W4 and W20 (new vaccination schedule).
  Interventions: Biological: Sm14 recombinant vaccine+ GLA-SE adjuvant

INTERVENTIONS:
Biological: Sm14 recombinant vaccine+ GLA-SE adjuvant — rSm14 - recombinant protein (GMP produced) - 50ug / injection GLA-SE- synthetic Glucopyranosyl lipid A in stable emulsion: 2.5ug / injection

SUMMARY:
Previous clinical trials have already demonstrated the safety of the candidate vaccine in adults as well as in children, in good health or infected with schistosomiasis. Regarding the induced immune response, more than 80% of vaccinated subjects were seroconverted after three vaccine injections. The induced immune response was substantial but transient. In order to obtain a more lasting immune response, the investigator will experiment with a new vaccination schedule (2 injections 1-month interval and the 3rd injection 5 months after the first dose), versus the vaccine schedule initially used (3 injections at 1-month interval).

This trial will be the last phase 2 before testing the efficacy of the rSm14 vaccine candidate.

DETAILED DESCRIPTION:
Adults with a history of infection with S. mansoni and / or S. haematobium, aged 18 to 49 years, pretreated with PZQ before the first vaccine injection (Inclusion) and living in villages in the Saint Louis region where schistosomiasis is endemic.

Comparative test with modification of the vaccine schedule previously used:

* The reference vaccine administration schedule consists of three vaccine administrations one-month interval (Group Vacc3).
* The new vaccine injection schedule will consist of a primary vaccination with two administrations of the vaccine one month apart, then a booster five (5) months after the first injection (Group Vacc2+1). Immunogenicity and safety will be evaluated and compared in these 2 groups.

These two groups of adults will be formed after randomization and pretreatment with PZQ (4 to 8 weeks before their first vaccine administration).

Main objective: to compare the immunological quality of the new vaccination schedule (amplitude and duration) versus the vaccination schedule used in the previous trials, by studying the Sm14 specific antibody response induced both quantitatively and qualitatively. The hypothesis is to obtain a mean response quantitatively higher with the new vaccine schedule.

Secondary objective: safety profile of the two vaccine schedules studied.

Regimen Group Vacc3 (reference group): Adults receiving 3 injections of the vaccine one month apart.

Group Vacc2+1 (experimental group): Adults receiving 2 injections of the vaccine one month apart then a third one five (5) months after the first injection.

Group Vacc3 : subjects will receive three (3) intramuscular injections into the deltoid muscle of 0.5mL of vaccine on Day 0, Week 4 and Week 8.

Group Vacc2+1 : subjects will receive three (3) intramuscular injections into the deltoid muscle of 0.5mL of vaccine on Day 0, Week 4 and Week 20.

Assessment of immunogenicity :

- Comparative Immunoassays between both groups: measures assessing differences in Sm14-specific antibody production several time points after third vaccine injection.

Antibody response evaluated on plasma obtained at:

* Time of the first dose
* 1 month after the third vaccine dose
* 3 months after the third vaccine dose
* 6 months after the third vaccine dose
* 9 months after the third vaccine dose Each subject will have 5 blood samples of 6mL, representing a total volume of 30 mL collected over the duration of the study.
* Cell markers and cytokines production Specific Sm14 cellular response (on PBMC) - production of intracellular cytokines and expression of specific immune markers - will be studied. A measure assessing change between two time points, i.e. time of the first dose and one month after the third injection of vaccine.

Assessment of Safety and Tolerance :

Emerging adverse events defined by an abnormal physical state or physical reaction that did not exist at baseline.

Emerging adverse events defined by abnormal variation in clinical constants. Emerging adverse events defined by abnormal levels of the serum products studied

Physical exams -

Physical exams includes :

Measurement of clinical constants

* Body temperature
* Respiratory rate at rest
* Heart rate at rest
* Blood pressure at rest (systolic + diastolic)

General examination

* Examination of the upper digestive tract (oral level)
* Abdominal examination
* Lung examination
* cardiovascular system examination

  * This will be carried out in the subjects preselected at the pre-inclusion visit, ie 8 days before inclusion.
  * And this will be carried out in subjects included in the clinical trial The physical exams will be carried out before each vaccine injection and followed by an observation at several post injection periods ie 1 hour, 2 hours, 24 hours and 48 hours.

After vaccination (following 3 vaccine injections) subjects will have a physical examination at 1, 3, 6 and 9 months after the third injection.

Thus, during the clinical trial, subjects after inclusion will have 9 medical exams.

Laboratory tests including :

* complete blood cell counts,
* hepatic function : dosage of serum transaminase (liver enzymes aspartate aminotransferase (AST) and alanine aminotransferase (ALT))
* renal function : serum creatinine
* serum albumin dosage These analyzes will be performed one week before inclusion (Vpi / W -1) to ensure that the subject is fit to receive the vaccine (satisfactory state of health).

Subsequently, and due to the excellent tolerance observed during previous clinical trials, a biological assessment will only be performed at the request of the investigators.

The villages identified for the clinical trial (n=3 or 4) will be selected approximately 3 months before subject inclusion. Only the adults having an infectious history will be considered for the subject selection.

No PZQ treatment is scheduled during the trial, however, if a person has a spontaneous complaint which is potentially symptomatic for schistosomiasis, parasitological testing will be performed. If the number of Sh eggs reaches 50 eggs / 10mL urine, and / or 400 EPG in stool for Sm, the subject will be treated. If the intensity of the infection is lower, the subject will not be treated but followed up regularly.

With the approval of the coordinator, the Investigator may decide to treat a subject at any time for security reasons.

At the end of the clinical trial, subjects will be tested for schistosomiasis and treated with PZQ if found positive.

Recruitment:

The villages identified for the clinical trial (n=3 or 4) will be selected approximately 3 months before subject inclusion. Only the adults having an infectious history will be considered for the subject selection.

Statistical consideration In terms of immunogenicity, the investigators expect to obtain induction of a significant anti-Sm14 specific immune response (Ab) in at least 70% of subjects (both groups combined). For group Vacc3, the residual average specific immune response one year after the first administration should be comparable to that obtained during phase 2a, ie 50% of the maximal response. For group Vacc2+1, the investigators expect a residual specific immune response at 1 year of 75%. So, an expected improvement in the immune response of 25%. Thus, for a statistical power fixed at 80%, an alpha risk at 5%, the number of subjects required using the Altmann nomogram method is 55 adults for each of the 2 groups.

Predicting a 10% loss to follow-up percentage, 120 subjects will be included in the clinical trial, or 60 subjects per group.

Duration Total duration of the study (32 months): November 2020 to July 2023 (inclusive).

Preparation phase (7-8 months; drafting of documents and submission); clinical trial (17 months (January-February 2022 to June-July 2023); post-trial, immunological analyzes and data management (6-7 months).

ELIGIBILITY:
Inclusion Criteria:

* Man living in villages in the Saint Louis region where schistosomiasis is endemic.
* Having an infectious history of schistosomiasis.
* Adult between 18 and 49 years old at the time of the first injection.
* Have received pre-treatment with PZQ four to eight weeks before inclusion.
* Consent signed by the volunteer after information.
* Satisfactory state of health, confirmed on clinical examination and following biological assessment (Vpi / W-1).
* Available for the duration of the trial.
* To be negative to the Covid-19 antigenic test

Exclusion Criteria (Non inclusion criteria) :

* Subject not meeting one of the inclusion criteria.
* Participation to a previous anti-schistosomiasis vaccine clinical trial.
* Participation in another ongoing clinical research
* Current or previous chronic administration (defined as more than 14 days) of immunosuppressive drugs or other immune modulating drugs.
* Known hypersensitivity to any component present in the Sm14 vaccine, or to any given vaccine, and / or history of allergic disease.
* Acute illness at the time of inclusion.
* Other conditions which, according to the PI, can potentially represent a danger to the subject to be included.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
assessment of Immunogenicity 1 | Day 1
  The anti-Sm14 IgG isotypes (Total IgG; IgG1; IgG3; IgG4; IgE) antibody response using an indirect ELISA
assessment of Immunogenicity 2 | Day 56
  The anti-Sm14 IgG isotypes (Total IgG; IgG1; IgG3; IgG4; IgE) antibody response using an indirect ELISA
assessment of Immunogenicity 3 | Day 84
  The anti-Sm14 IgG isotypes (Total IgG; IgG1; IgG3; IgG4; IgE) antibody response using an indirect ELISA
assessment of Immunogenicity 4 | Day 140
  The anti-Sm14 IgG isotypes (Total IgG; IgG1; IgG3; IgG4; IgE) antibody response using an indirect ELISA
assessment of Immunogenicity 5 | Day 168
  The anti-Sm14 IgG isotypes (Total IgG; IgG1; IgG3; IgG4; IgE) antibody response using an indirect ELISA
assessment of Immunogenicity 6 | Day 224
  The anti-Sm14 IgG isotypes (Total IgG; IgG1; IgG3; IgG4; IgE) antibody response using an indirect ELISA
assessment of Immunogenicity 7 | Day 308
  The anti-Sm14 IgG isotypes (Total IgG; IgG1; IgG3; IgG4; IgE) antibody response using an indirect ELISA
assessment of Immunogenicity 8 | Day 392
  The anti-Sm14 IgG isotypes (Total IgG; IgG1; IgG3; IgG4; IgE) antibody response using an indirect ELISA
assessment of immunogenicity 9 | Day 1
  Measure expression change in membrane markers expression of PBMC under in vitro Sm14 antigen activation
assessment of immunogenicity 10 | Day 84
  Measure expression change in membrane markers expression of PBMC under in vitro Sm14 antigen activation (for Group Vacc3)
assessment of immunogenicity 11 | Day 168
  Measure expression change in membrane markers expression of PBMC under in vitro Sm14 antigen activation (for Group Vacc2+1)
assessment of immunogenicity 12 | Day 1
  12. Measure cytokine production (ELISA) by PBMC under in vitro Sm14 antigen activation
assessment of immunogenicity 13 | Day 84
  12. Measure cytokine production (ELISA) by PBMC under in vitro Sm14 antigen activation (for Group Vacc3)
assessment of immunogenicity 14 | Day 168
  12. Measure cytokine production (ELISA) by PBMC under in vitro Sm14 antigen activation (for Group Vacc2+1)

SECONDARY OUTCOMES:
Safety of the vaccine candidate Sm14 -1 | from Day 1 to Day 442
  The occurrence of study vaccine-related SAEs
Safety of the vaccine candidate Sm14 - 2 | from Day 1 to Day 3
  2. The occurrence of solicited injection site reactogenicity
Safety of the vaccine candidate Sm14 -3 | from Day 28 to Day 30
  The occurrence of solicited injection site reactogenicity
Safety of the vaccine candidate Sm14 -4 | from Day 56 to Day 58
  The occurrence of solicited injection site reactogenicity for Group Vacc3
Safety of the vaccine candidate Sm14 -5 | from Day 140 to Day 142
  The occurrence of solicited injection site reactogenicity for Group Vacc2+1
Safety of the vaccine candidate Sm14 _6 | from Day 1 to Day 3
  The occurrence of solicited injection site reactogenicity
Safety of the vaccine candidate Sm14 -7 | from Day 28 to Day 30
  The occurrence of solicited injection site reactogenicity
Safety of the vaccine candidate Sm14 -8 | from Day 56 to Day 58
  The occurrence of solicited injection site reactogenicity for Group Vacc3
Safety of the vaccine candidate Sm14 -9 | from Day 140 to Day 142
  The occurrence of solicited injection site reactogenicity for Group Vacc2+1

CONTACTS AND LOCATIONS:
Overall Officials: Gilles RIVEAU, PharmD PhD, Study Director — Biomedical Research Center EPLS
Locations (1):
- Biomedical Research Center EPLS, Saint-Louis, Senegal

IPD SHARING:
Plan to Share IPD: No